CLINICAL TRIAL: NCT02674646
Title: RandOmized Study Exploring the Combination of radioTherapy With Two Types of Acupuncture Treatment: The ROSETTA Trial
Acronym: ROSETTA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Stephanie Combs, Univ.-Prof. Dr. med., Professor and Chair, Radiation Oncology, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ROSETTA
Record Dates: First submitted 2015-12-08; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Verum Acupuncture (Experimental): Group A: Verum Acupuncture (Needle Acupuncture) Needlepoints Bilateral PC 6, S 36, L 8, L 9 Unilateral R4, R 6 Acupuncture will be applied for approx. 20 min. with 10 needlepoints. Standard radiotherapy
  Interventions: Radiation: Radiotherapy; Device: Needle Acupuncture
- Group B: Sham Acupuncture (Sham Comparator): Group B: Sham Acupuncture (Needle Acupuncture) Needlepoints 8 needles in the medioaxillary line below the 6th rib, bilateral 2 needles unilateral Sham-acupuncture will be applied for approx. 20 min. with 10 needlepoints. Standard radiotherapy
  Interventions: Radiation: Radiotherapy; Device: Needle Acupuncture

INTERVENTIONS:
Radiation: Radiotherapy — Radiation as indicated by the cancer diagnosis
Device: Needle Acupuncture — Needle Acupuncture according to Traditional Chinese Medicine (TCM)

SUMMARY:
The ROSETTA-trial will evaluate the effect of acupuncture as a complementary treatment parallel to radiation therapy in oncological patients. The trial is designed as a two-armed trial. Depending on the treatment study arm either verum- or Sham sham-acupuncture will be applied. Acupuncture is applied treatment bi-weekly during the first week of radiotherapy, thereafter weekly until the end of radiotherapy; the follow-up visits include clinical workup as well as questionnaires.

DETAILED DESCRIPTION:
Adverse effects such as fatigue, pain, skin problems , nausea and vomiting are commonly known in patients undergoing irradiation alone or in combination with chemotherapy (RCHT). Patients suffering from these symptoms are constricted severely in their daily life and their quality of life (QOL) is often reduced. As examined several times, acupuncture can cause an amelioration of these specific disorders. Especially for pain symptoms several groups have shown efficacy of acupuncture. To what extent a difference between traditional acupuncture (verum-acupuncture) and false acupuncture (sham-acupuncture) can cause reduction of side effects and improvement of QOL is not clarified. Therefore, the ROSETTA trial is a randomized trial with two treatment arms.

The verum-group receives "real acupuncture" , while the Sham-group is treated with sham- acupuncture points. These points are "nonsense" needlepoints, which do not have any correlate in TCM.

Patients are going to get standardized questionnaires (EORTC QOL C-30) before their first, after their fourth and after their last acupuncture treatment. Patients will be questioned about their condition by the investigator. The answers will be documented according to the standardized scoring system CTCAE (Common Toxicity Criteria for Adverse Events).

Group A: Verum Acupuncture Needlepoints Bilateral PC 6, S 36, L 8, L 9 Unilateral R4, R 6

Group B: Sham Acupuncture Needlepoints 8 needles in the medioaxillary line below the 6th rib, bilateral 2 needles unilateral

ELIGIBILITY:
Inclusion Criteria

Patients meeting all of the following criteria will be considered for admission to the trial:

* treatment with radiotherapy
* age ≥ 18 years of age
* Ability ability of subject to understand character and individual consequences of the clinical trial
* written informed consent (must be available before enrolment in the trial)

Exclusion Criteria

Patients presenting with any of the following criteria will not be included in the trial:

* any contraindication to acupuncture
* known coagulopathy or anticoagulation therapy with bleeding time > 4 minutes, thrombocyte count < 50 000/μl
* missing compliance
* skin disease in the region of the acupuncture points
* refusal of the patients to take part in the study
* participation in another clinical study or observation period of competing trials,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 6 weeks after completion of radiotherapy
  questionnaire

SECONDARY OUTCOMES:
Fatigue | 6 weeks after radiotherapy
  Fatigue measures by questionnaire and fatigue scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Combs, Prof. Dr., Principal Investigator — Klinikum rechts der Isar, Radiation Oncology, Professor and Chair

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asadpour R, Kessel KA, Bruckner T, Sertel S, Combs SE. Randomized study exploring the combination of radiotherapy with two types of acupuncture treatment (ROSETTA): study protocol for a randomized controlled trial. Trials. 2017 Aug 29;18(1):398. doi: 10.1186/s13063-017-2139-5. PMID 28851420